CLINICAL TRIAL: NCT01161082
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending Single to Multi-Dose Study of Safety, Tolerability, and Bioeffect of Subcutaneously Administered REGN727 in Patients With and Without Concomitant Atorvastatin
Brief Title: Ascending Multi-dose Study of REGN727(SAR236553) With and Without Concomitant Atorvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R727-CL-1001
Record Dates: First submitted 2010-07-09; First posted 2010-07-13 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2011-11

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Group 1 with atorvastatin (Experimental): Dose 1 versus placebo
  Interventions: Drug: REGN727(SAR236553)
- Group 2 with atorvastatin (Experimental): Dose 1 versus placebo
  Interventions: Drug: REGN727(SAR236553)
- Group 3 with atorvastatin (Experimental): Dose 2 versus placebo
  Interventions: Drug: REGN727(SAR236553)
- Group 4 with atorvastatin (Experimental): Dose 2 versus placebo
  Interventions: Drug: REGN727(SAR236553)
- Group 5 with atorvastatin (Experimental): Dose 3 versus placebo
  Interventions: Drug: REGN727(SAR236553)
- Group 6 with atorvastatin (Experimental): Dose 3 versus placebo
  Interventions: Drug: REGN727(SAR236553)
- Group 7 without atorvastatin (Experimental): Dose 3 versus placebo
  Interventions: Drug: REGN727(SAR236553)
- Group 8 with atorvastatin (Experimental): Dose4 versus placebo
  Interventions: Drug: REGN727(SAR236553)

INTERVENTIONS:
Drug: REGN727(SAR236553) — subcutaneous

SUMMARY:
This study will test the safety, tolerability, and bioeffects (how the body reacts to the drug) of REGN727 compared with placebo (an inactive substance that contains no medicine) in hyperlipidemic patients with or without atorvastatin therapy. The study drug and placebo will be administered by subcutaneous injection at the clinic. There will be a total of 2 or 3 study drug injections over 16 clinic visits, which will include 3 overnight stays(study duration 148 days, not including the screening period). Patients on atorvastatin will take their daily dose in the morning for the duration of the study. Patients will be monitored by the study staff for side effects and the body's response to the study drug. Vital signs(blood pressure, temperature, breathing and heart rate) will be checked, and blood and urine samples will be collected at some or all visits.

ELIGIBILITY:
Inclusion Criteria

* Men and women with elevated cholesterol on stable doses of atorvastatin 10-40mg/day regimen
* Body mass index between 18.0 and 35.0 kg/m2, inclusive
* For women of childbearing potential, a negative serum pregnancy test at the screening visit and a negative urine pregnancy test on day -2 or day -1
* For men and women of childbearing potential, willingness to utilize adequate contraception and not become pregnant (or have their partner[s] become pregnant)during the full duration of the study
* Willing, committed and able to return for all the clinic visits and complete all study-related procedures
* Able to read, and able to sign the informed consent form

Exclusion Criteria:

* History of MI, ACS, Angina, Stroke, peripheral vascular disease, or cardiac revascularization
* Pregnant or breast-feeding women
* Blood donation of any volume within 1 month prior to administration of study drug
* Congestive heart failure
* Consumption of greater than 1 quart of grapefruit juice per day
* Previous exposure to any therapeutic or investigational biological agent within 30 days of screening
* History of alcohol or drug abuse within one year to the screening visit

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint in the study is to assess the incidence and severity of treatment-emergent adverse events in hyperlipidemic patients treated with REGN727 or placebo receiving stable doses of atorvastatin. | visit 4 (day 1) to visit 16 (day 148)

SECONDARY OUTCOMES:
To assess the pharmacodynamic effect of REGN727 added to atorvastatin on lipids | Visit 4 (Day 1) to Visit 16 (Day 148)
To assess the pharmacodynamic effect of monotherapy REGN727 in hyperlipidemic patients | Visit 4 (Day 1) to Visit 16 (Day 148)
To assess the pharmacokinetics of REGN727 in hyperlipidemic patients with or without atorvastatin | Visit 4 (Day 1) to Visit 16 (Day 148)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Swergold, MD, PhD, Study Director — Regeneron Pharmaceuticals
Locations (2):
- United States (2):
  - Site 1, Cincinnati, Ohio
  - Site 2, Knoxville, Tennessee

REFERENCES:
- [Derived] Stein EA, Mellis S, Yancopoulos GD, Stahl N, Logan D, Smith WB, Lisbon E, Gutierrez M, Webb C, Wu R, Du Y, Kranz T, Gasparino E, Swergold GD. Effect of a monoclonal antibody to PCSK9 on LDL cholesterol. N Engl J Med. 2012 Mar 22;366(12):1108-18. doi: 10.1056/NEJMoa1105803. PMID 22435370